CLINICAL TRIAL: NCT00449839
Title: Changes of the Infusion Rate in Insulin Pump Treatment. A Randomized, Unblinded Cross-Over Study.
Brief Title: Changes of the Infusion Rate in Insulin Pump Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Jens Sandahl Christiansen, Prof.Dr.Med, Aarhus University Hospital, department of Endocrinology and Diabetes
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDS 265 PK IAsp 2006/199
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes
Keywords: Insulin pump treatment CSII; Absorption; Insulin Aspart
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A, CSII without bolus (Other): Period A: A constant subcutaneous infusion rate of insulin aspart (0.5 U/hr) is given for 8 hours. Following 3 hours of blood sampling.
  Interventions: Drug: Insulin Aspart
- B; CSII with bolus (Other): Period B: A constant subcutaneous infusion of insulin aspart (0.5 U/hr) is given for 8 hours and upon start a s.c.bolus (1.4 U)of insulin aspart is given. Hereafter follows 3 hours of blood sampling.
  Interventions: Drug: Insulin Aspart
- C; CSII with bolus, optional (Other): A constant subcutaneous insulin aspart infusion is given for 8 hours and upon start a bolus of insulin aspart is given. The bolus in arm C is of a different size then arm B. After the 8 hours of constant infusion follows 3 hours of blood sampling. Period C are optional and it is evaluated if it will be conducted after period A and B has been performed.
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Aspart — A; CSII without bolus: 8 hours of constant insulin infusion. B; CSII with bolus: 8 hours of a constant insulin infusion starting with a s.c. bolus.
  C; CSII with bolus, optional: 8 hours of a constant insulin infusion starting with a different bolus than period B. This period is optional and it will be evaluated after period A and B if period C is conducted.
  Other Names: Insulin Aspart/NovoRapid

SUMMARY:
A pharmacokinetic study of insulin pump treatment using Insulin Aspart. The study consist of three different periods A, B and C where a constant the insulin infusion rate is given during the periods. In period B and C will the infusion start with a bolus.

It will be investigated if a steady state of insulin will be obtained faster in period B and C then A.

DETAILED DESCRIPTION:
A pharmacokinetic study of insulin pump treatment using Insulin Aspart. The study consist of three different periods A, B and C where a constant the insulin infusion rate is given during the periods. Each period will last 12 hours and blood will be drawn to measure absorbed Insulin Aspart. During period A will a constant the infusion rate of insulin be given. In period B and C will there at the start of the constant infusion rate be given a bolus. The bolus in period C is calculated on the basis of the results in period B, therefore will all participants experience period C last where as period A and B is randomized cross-over. Period C is written in the protocol as optional and it is evaluated after period A and B if period C will be performed.

The hypothesis is that steady state of insulin will be obtained faster in period B and C than A.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Healthy volunteer
* Men and women between ≥18 and <50 years
* Women in the child-bearing age should be sufficient protected against pregnancy (use birth control pill or intrauterine device or be sterilized or hysterectomized)
* BMI between 18-30 kg/m^2 (both included)

Exclusion Criteria:

* Suspected or known allergy against the drug used in the study or similar drugs
* Previous history of endocrinology disease (including Diabetes Mellitus)
* Suspected or known alcohol- or drug abuse
* Any disease influencing the study, evaluated by the investigator
* Pregnancy, breast-feeding or the wish of becoming pregnant during the study period. Furthermore women in the child bearing age not sufficient protected against pregnancy (sufficient is: use of birth control pill or intrauterine device or be sterilized or hysterectomized)
* Participation in other research projects during the last 3 months before this project

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Absorbed Insulin Aspart | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sandahl Christiansen, Prof. Dr.Med, Principal Investigator — Aarhus University Hospital, department of Endocrinology and Diabetes
Locations (1):
- Aarhus University Hospital, department of Endocrinology and Diabetes, Aarhus C, Aarhus, Denmark